CLINICAL TRIAL: NCT02104999
Title: Technical Accuracy and Userfriendliness of a Point-Of-Care C Reactive Protein (CRP) Device in Comparison With Laboratory CRP Testing in Nursing Home Residents.
Brief Title: Technical Accuracy and Userfriendliness of a Point-Of-Care C Reactive Protein Device in a Nursing Home Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Latour Katrien, Research Assistant, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRP-NH0414
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Older Adults; Ill Older Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Point-of-care test for CRP (Other): Device: C Reactive Protein (CRP) measurement on capillary blood using a point-of-care test to determine the CRP level in the blood
  Interventions: Device: Point-of-care test for CRP

INTERVENTIONS:
Device: Point-of-care test for CRP — Device: C Reactive Protein (CRP) measurement on capillary blood using a point-of-care test to determine the CRP level in the blood

SUMMARY:
Study to test the technical accuracy and userfriendliness of a Point-of-care C Reactive Protein device (POC CRP device) in comparison with laboratory CRP testing in nursing home residents

ELIGIBILITY:
Inclusion Criteria:

* Older (65 years or older) nursing home residents

Exclusion Criteria:

* Residents not understanding Dutch

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Technical accuracy | 2 month
  Correlation between the results of the Point-of-care C Reactive Protein device and the results of the laboratory

SECONDARY OUTCOMES:
User-friendliness | 2 months
  Evaluation of the user-friendliness on a five point Likert-scale. Following items are scored: device start-up, test duration, sample size, test characteristics, calibration, measuring range, handling of test tubes, filling of the capillary, placing the test cartridge, test recording and additional material usage.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Buntinx, PhD, Principal Investigator — KU Leuven
Locations (1):
- Domino vzw, Ghent, Oost-Vlaanderen, Belgium